CLINICAL TRIAL: NCT00104767
Title: A Phase I Trial to Evaluate Cyclooxygenase 2 Inhibitor-Mediated Modulation of T Regulatory Cells in Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Celecoxib in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000415733; UCLA-0407028-01; NCT00744783 (obsolete NCT alias)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- celecoxib (Experimental)
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: celecoxib

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also stimulate the immune system in different ways and stop tumor cells from growing.

PURPOSE: This phase I trial is studying the side effects and best dose of celecoxib in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the optimal biologic dose (OBD) of celecoxib that is necessary to decrease peripheral blood lymphocyte CD4+ and CD25+ T-lymphocyte regulatory cells in patients with stage IIIB or IV non-small cell lung cancer.

Secondary

* Determine the OBD of this drug that is necessary to decrease peripheral blood lymphocyte FOXP3 levels in these patients.

OUTLINE: This is a nonrandomized, dose-escalation study.

Patients receive oral celecoxib twice daily on days 1-7 in the absence of unacceptable toxicity.

Cohorts of 3 patients receive escalating doses of celecoxib until the optimal biologic dose (OBD) is determined. The OBD is defined as the lowest dose that results in the maximum decrease in peripheral blood lymphocyte CD4+ and CD25+ T-lymphocyte regulatory cells and FOXP3 levels where no dose-limiting toxicity occurs. An additional 15 patients are treated at the OBD.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer
* Stage IIIB or IV disease
* Radiographically measurable disease
* 18 and over
* Performance status: ECOG 0-2
* Renal: Creatinine ≤ 2 mg/dL
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 4 weeks since prior chemotherapy
* Endocrine therapy: More than 4 weeks since prior corticosteroids; No concurrent corticosteroids, including chronic corticosteroids, except for medically-indicated topical steroids
* Radiotherapy: More than 4 weeks since prior radiotherapy
* More than 4 weeks since other prior anticancer therapy
* More than 4 weeks since prior non-cytotoxic investigational agents
* At least 72 hours since prior nonsteroidal anti-inflammatory drugs (NSAIDs)

Exclusion Criteria:

* pregnant or nursing
* comorbid disease, psychiatric condition, chronic medical condition, or laboratory abnormality that would preclude study treatment or compliance with study requirements
* hypersensitivity to celecoxib, sulfonamides, aspirin, other NSAIDs, or any study reagent
* history of gastrointestinal ulceration, bleeding, or perforation
* other concurrent cyclooxygenase-2 or -3 inhibitors
* other concurrent NSAIDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-01; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Optimal biologic dose (OBD) necessary to decrease peripheral blood lymphocyte (PBL) CD4+ and CD25+ T-lymphocyte regulatory cells at 1 week | 7 days

SECONDARY OUTCOMES:
OBD necessary to decrease PBL FOXP3 levels at 1 week | 7 dayd
Function of CD4+ and CD25+ T-regulatory cells at 1 week | 7 days
Markers of cyclooxygenase-2 (COX-2) dependent gene expression before and after treatment at 1 week | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garon, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States